CLINICAL TRIAL: NCT01971684
Title: ICON1: Physician Treatment Decisions and Patient-Reported Outcomes in Pediatric Refractory Immune Thrombocytopenia
Brief Title: ICON1: Treatment Decisions and Outcomes in Pediatric Refractory ITP
Acronym: ICON1
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Terrana ITP Research Fund (Other)
Responsible Party: Principal Investigator, Rachael Grace, Principal Investigator, PKD Natural History Study, Boston Children's Hospital
Other Study IDs: P00008709
Record Dates: First submitted 2013-10-21; First posted 2013-10-29 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP; idiopathic thrombocytopenic purpura; bleeding score; platelet count; health-related quality of life; HRQL; Purpura; Purpura, Thrombocytopenic; Purpura, Thrombocytopenic, Idiopathic; Blood Coagulation Disorders; Hematologic Diseases; Hemorrhage; Skin Manifestations; Thrombocytopenia; Blood Platelet Disorders; Immune System Diseases; Hemorrhagic Disorders; Autoimmune Diseases; Therapeutic Uses
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Purpura; Purpura, Thrombocytopenic; Blood Coagulation Disorders; Hematologic Diseases; Hemorrhage; Skin Manifestations; Thrombocytopenia; Blood Platelet Disorders; Immune System Diseases; Hemorrhagic Disorders; Autoimmune Diseases | interventions — Rituximab; Mercaptopurine; Mycophenolic Acid; Sirolimus; Splenectomy; romiplostim; eltrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Refractory Pediatric ITP Patients: Pediatric ITP patients, ages 1-18, starting a new second line ITP therapy, defined as not IVIG, steroids, anti-D, or aminocaproic acid.
  Interventions: Drug: Second Line ITP agents

INTERVENTIONS:
Drug: Second Line ITP agents — The treating physicians will select the second line agent and clinical data will be collected.
  Other Names: rituximab; 6-mercaptopurine; mycophenolate mofetil; sirolimus; splenectomy; romiplostim; eltrombopag

SUMMARY:
The purpose of this study is to understand physician treatment decisions in selecting specific second line treatments in pediatric ITP and to determine the effectiveness of different second line ITP treatments. Eligible patients are those ages 1-18 years who are starting on a new second line treatment for ITP, defined as any treatment other than IVIG, steroids, anti-D globulin, or aminocaproic acid. Enrolled patients remain on the study for approximately one year.

DETAILED DESCRIPTION:
The purpose of this observational study is to model factors that determine physician treatment decisions in selecting specific second line agents in pediatric ITP and to determine the comparative effectiveness of second line ITP treatments by bleeding measures, platelet counts, and patient reported outcome measures. This prospective observational, longitudinal, multicenter cohort study will aim to collect routine clinical care data, quality of life information from patients, and decision making data from clinicians at enrollment and at regular clinical intervals for at least one year. The primary and secondary objectives are as follows:

Primary Objectives:

1. To model factors that determine physician treatment decisions in selecting specific second line agents in pediatric ITP.
2. To assess patient reported outcomes with relation to specific second line pediatric ITP therapies.
3. To determine the comparative effectiveness of second line ITP treatments in terms of bleeding and platelet counts.

Secondary Objectives:

1. To describe phenotypic variation among patients with refractory ITP;
2. To assess side effects and complications related to specific treatments for refractory ITP;
3. To describe monitoring and follow up practices among pediatric hematologists with each second line agent;
4. To weight factors that physicians use when deciding to treat pediatric ITP patients with second line agents;
5. To determine whether physician perception of patient quality of life correlates with patient derived quality of life measures;
6. To measure the correlation between the ITP Bleeding Scale and the Bleeding Assessment Tool in refractory pediatric ITP patients.

ELIGIBILITY:
Inclusion Criteria:

* Immune Thrombocytopenia or Evans Syndrome
* Ages > 12 months to <18 years
* Starting a new second line therapy as defined as any therapy except IVIG, steroids, anti-D globulin, or aminocaproic acid
* Starting a single agent/monotherapy

Exclusion Criteria:

* Evans Syndrome with a history of or current evidence of autoimmune hemolytic anemia
* Unwillingness to be followed for 1 year
* Physician providing care is unwilling to participate
* Patient is starting multiple second line agents simultaneously

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric refractory ITP patients starting on a new second line therapy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
change from baseline in patient reported outcomes | Enrollment, 1 and 12 months
  Kids ITP Tool, Memorial Symptom Assessment Scale, Fatigue Scale
change from baseline in bleeding assessment | Enrollment, 1, 6, and 12 months
  ITP Bleeding Scale, Bleeding Assessment Tool
change from baseline in platelet count | over 1 year

SECONDARY OUTCOMES:
side effects and complications of treatments | 1 year

CONTACTS AND LOCATIONS:
Locations (29):
- United States (26):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Mattel Children's Hospital, Los Angeles, California
  - Children's Hospital of Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - UCSF School of Medicine, San Francisco, California
  - Colorado Children's Hospital, Denver, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - St. John Hospital & Medical Center, Detroit, Michigan
  - Goryeb Children's Hospital, Morristown, New Jersey
  - Columbia University Medical Center, New York, New York
  - New York-Presbyterian University Hospital of Columbia and Cornell, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - St. Jude's Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's, Seattle, Washington
- Canada (3):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - U. de Montreal CHU St. Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grace RF, Shimano KA, Bhat R, Neunert C, Bussel JB, Klaassen RJ, Lambert MP, Rothman JA, Breakey VR, Hege K, Bennett CM, Rose MJ, Haley KM, Buchanan GR, Geddis A, Lorenzana A, Jeng M, Pastore YD, Crary SE, Neier M, Neufeld EJ, Neu N, Forbes PW, Despotovic JM. Second-line treatments in children with immune thrombocytopenia: Effect on platelet count and patient-centered outcomes. Am J Hematol. 2019 Jul;94(7):741-750. doi: 10.1002/ajh.25479. Epub 2019 Apr 29. PMID 30945320
- [Result] Grace RF, Despotovic JM, Bennett CM, Bussel JB, Neier M, Neunert C, Crary SE, Pastore YD, Klaassen RJ, Rothman JA, Hege K, Breakey VR, Rose MJ, Shimano KA, Buchanan GR, Geddis A, Haley KM, Lorenzana A, Thompson A, Jeng M, Neufeld EJ, Brown T, Forbes PW, Lambert MP. Physician decision making in selection of second-line treatments in immune thrombocytopenia in children. Am J Hematol. 2018 Jul;93(7):882-888. doi: 10.1002/ajh.25110. Epub 2018 May 6. PMID 29659042